CLINICAL TRIAL: NCT04581759
Title: Endovascular Treatment Combined With Remote Ischemic Postconditioning in Patients With Acute Ischemic Stroke Improves the Prognosis，a Multicenter, Randomized, Prospective Trial
Brief Title: Endovascular Treatment and RIPC in Acute Ischemic Stroke
Acronym: EnTRIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); Shaanxi Provincial People's Hospital (Other); Xijing Hospital (Other); Tang-Du Hospital (Other); Xi'an No.3 Hospital (Other Government); Xi'an Gaoxin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2020-015
Record Dates: First submitted 2020-09-09; First posted 2020-10-09 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Acute Ischemic Stroke; Endovascular Treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC (Experimental): Patients in the RIPC group not only receive foundational treatment but also have five cycles of 5-min cuff inflation followed by 3-min deflation to the bilateral upper arm using a RIPC device (IPC-906X; Beijing Renqiao Institute of Neuroscience, Beijing, China) after endovascular treatment while in-hospital.
  Interventions: Device: RIPC device (IPC-906X); Drug: foundational treatment
- foundational treatment group (FT) (Sham Comparator): Patients in the FT group only receive foundational treatment, including free radical elimination in the acute stage, blood pressure and blood glucose stabilization, and antiplatelet (aspirin or/and clopidogrel,100-300mg/d) and lipid-lowering (atorvastatin 20-60mg/d,rosuvastatin 10-20mg/d) drugs, during the study period without remote ischemic postconditioning after endovascular treatment.
  Interventions: Drug: foundational treatment

INTERVENTIONS:
Device: RIPC device (IPC-906X) — Patients in the RIPC group will have five cycles of 5-min cuff inflation followed by 3-min deflation to the bilateral upper arm twice a day after Mechanical Thrombectomy.
  Arms: RIPC
Drug: foundational treatment — foundational treatment, including free radical elimination in the acute stage, blood pressure and blood glucose stabilization, and antiplatelet (aspirin or/and clopidogrel ) and lipid-lowering (statins) drugs

SUMMARY:
Endovascular treatment（ET）is an effective therapy for acute ischemic stroke(AIS) with great vessel obstruction. However, acute complications such as high postoperative perfusion injury, hemorrhagic transformation and restenosis resulted in functional independence in only about 50% of patients 90 days after interventional surgery. Therefore, it is very important to protect the neurologic function after emergency endovascular treatment. The investigators' previous studies have shown that combined with intravenous thrombolytic therapy and remote postconditioning（RIPC）can significantly improve the neurological impairment and short-term and long-term prognosis in patients with acute stroke. In this multicenter, randomized controlled trial, the investigators assumed patients with acute ischemic stroke who had successfully revascularization after ET might benefit from RIPC as well. Patients in the RIPC group had five cycles of 5-min cuff inflation followed by 3-min deflation to the bilateral upper arm after ET. The primary endpoint measure was the proportion of patients with a favorable recovery of nerve function deficient assessed by Modified Rankin Scale （mRS≤2） 90 days after surgery. Secondary endpoints included the following: (1) Symptom endpoints: Neurological intelligence and function scores, postoperative hemorrhagic transformation rate, etc. (2) Blood index test: postoperative inflammatory factors, neuron-specific enolase (NSE) and other indicators. (3) Imaging endpoints: MRI-FLAIR , TCD, etc.

ELIGIBILITY:
Inclusion Criteria:

1. acute ischemic stroke（AIS） patients with large vessel occlusion (internal carotid artery system and vertebral basilar artery system) within 24 hours after onset, endovascular treatment (mechanical thrombotomy, intra-arterial thrombolysis, balloon dilatation or stent angioplastyand) successful opening were performed, and the definition of successful opening was defined by Modified Thrombolysis standard [Modified Thrombolysis in Cerebral infarction, mTICI]≥ 2B，The standards of endovascular interventional treatment are in line with the indications and contraindications formulated in the Chinese Guidelines for the Early Treatment of Acute Ischemic Stroke 2018；
2. Modified Rankin scale score (mRS) ≤1 before onset:
3. The Alberta Stroke Program Early CT score (ASPECTS)≥6 on admission;
4. National Institute of Health Stroke Scale (NIHSS) score ≥6 on admission;
5. Provision of written informed consent.

Exclusion Criteria:

1. CT or MRI scan showed significant midline deviation and the mass effect;
2. Glasgow(GCS) score ≤8 on admission;
3. failure to accomplish 3-months and 6-months follow up;
4. Severe cardiac, liver, or kidney disease, malignancy, severe coagulation dysfunction, severe anemia and systemic organ dysfunction;
5. Pregnant or nursing women, or patients with moderate to severe mental disorders or dementia;
6. Severe soft tissue injuries, fractures, thrombosis and other known peripheral vascular lesions of the upper limbs，active visceral hemorrhage, acute stage of fundus hemorrhage, cerebral aneurysm or cerebral arteriovenous malformation, and other unsuitable for bilateral upper arm compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale (mRS) | 7days, 90 days and 180 days after the surgery and at discharge
  The percentage of patients with a favorable outcome from baseline at 90 days and 180 days postoperatively, defined as a score of 0 or 2 on the modified Rankin scale (mRS)（Notes:mRS score from 0-6, higher scores mean worse outcome）

SECONDARY OUTCOMES:
The change of NIHSS score | 7days, 90 days and 180 days after the surgery and at discharge
  The percentage of functional recovery from baseline at 90 days and 180 days postoperatively, as measured by the National Institute of Health Stroke Scale, short for NIHSS（Notes:NIHSS score from 0-42. higher scores mean worse outcome）
The change of Barthel Index | 7days, 90 days and 180 days after the surgery and at discharge
  The change of functional recovery from baseline at 90 days and 180 days postoperatively, as measured by the Barthel Index （Notes:Barthel Index score from 0-100. higher scores mean better outcome）
The change of Montreal Cognitive Assessment (MoCA) score | 7days, 90 days and 180 days after the surgery and at discharge
  The change of cognitive recovery from baseline at 90 days and 180 days postoperatively, as measured by the MoCA （Notes:MoCA score from 0-30. higher scores mean better outcome）
The change of MMSE score | 7days, 90 days and 180 days after the surgery and at discharge
  The change of cognitive recovery from baseline at 90 days and 180 days postoperatively, as measured by the MMSE（Notes:MMSE score from 0-30. higher scores mean better outcome）
The change of inflammatory indicators | before ET, 24 hours and 7 days after the surgery
  Peripheral venous blood was drawn before Endovascular Treatment(ET) and 24 hours and 7 days postoperatively to determine the effect of repeated RIPC on anti-inflammatory (hIL-1β、hIL-2R、hIL-6、hIL8、hIL-10、S100-β、TNF-α) （Notes: unit ng/ml）
The change of angiogenic factors | before ET, 24 hours and 7 days after the surgery
  Peripheral venous blood was drawn before ET and 24 hours and 7 days postoperatively to determine the effect of repeated RIPC on vascular (VEGF、bFGF、EPO、HIF-1α、BDNF) and other pathways (S100B、NSE)（Notes: unit ng/ml）
The change of hemoglobin and Blood viscosity | up to 7 days after the surgery
  Peripheral venous blood was drawn before ET and 24 hours and 7 days postoperatively to determine the effect of repeated RIPC on Hb and Blood viscosity（Notes: unit g/L , mPa.s）
Postoperative hemorrhagic transformation | 72 hours after ET and hospitalization
  The proportion of patients with postoperative hemorrhagic transformation, based on CT scan and symptom
The change of MRI FLAIR Fazekas score | the changs from within 7 days to 90 days after the surgery
  Cerebral white matter demyelination measured by MRI FLAIR Fazekas score，（Notes:Fazekas score from 0-6. higher scores mean worse outcome）
The change of blood flow velocity | the changs from 24 hours after ET to 7 days after the surgery
  Vascular blood flow velocity measured by transcranial doppler （TCD） examination
Vascular resistance | the changs from 24 hours after ET to 7 days after the surgery
  Vascular resistance measured by TCD examination
mortality rate | up to 90 days and 180 days
  90-days and 180-days mortality rate
recurrence rate of cerebrovascular disease | up to 90 days and 180 days
  90-days and 180-days recurrence rate of cerebrovascular disease
blood pressure | up to 7days
  The effect of RIPC on blood pressure
heart rate | up to 7days
  The effect of RIPC on heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12/31/2023, for 1 year